CLINICAL TRIAL: NCT02772861
Title: Randomised Cross-over Single-site Study on the Bioavailability of Citrulline After an Oral Bolus of Citrulline, Glutamine, Arginine, 3-Methylhistidine or Placebo in Healthy Subjects
Brief Title: Citrulline Challenge Study for Healthy Subjects in the United Kingdom
Acronym: CHS-UK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 10/0458
Record Dates: First submitted 2011-12-05; First posted 2016-05-16 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-05

CONDITIONS: Intestinal Diseases
MeSH Terms: conditions — Intestinal Diseases | interventions — 3-methylhistidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Citrulline (Experimental): Citrulline is a non-protein amino acid that is present in substantial amounts in watermelon (Citrullus vulgaris), with a mean content of 2.1 mg/g fresh weight, ranging from 0.5 to 3.6 mg/g according to variety. The oral dose can reach 20 g, which was administered orally in the present study in one single dose, followed by a washout period of one week Amino Acid Supplement - One dose
  Interventions: Dietary Supplement: Amino Acid Supplement - One dose
- Glutamine (Experimental): L-glutamine is a protein amino acid found in proteins of all life forms. It is classified as a semi-essential or conditionally essential amino acid. This means that under normal circumstances the body can synthesize sufficient l-glutamine to meet physiological demands. However, there are conditions where the body cannot do so. Recently, l-glutamine has come to be regarded as one of the most important of the amino acids when the body is subjected to such metabolic stress situations as trauma (including surgical trauma), cancer, sepsis and burns. In the present study, glutamine was administered orally in one single dose of 20 g, followed by a washout period of one week.
  Amino Acid Supplement - One dose
  Interventions: Dietary Supplement: Amino Acid Supplement - One dose
- Arginine (Experimental): Arginine was administered orally in 20 g for one single dose, followed by a washout period of 1 week.
  Amino Acid Supplement - One dose
  Interventions: Dietary Supplement: Amino Acid Supplement - One dose
- 3-Methyl-Histidine (Experimental): This amino acid is made by methylation of the actin and myosin peptide chains in the muscle. Metabolism after intravenous administration of L-3-methylhistidine involves excretion in the urine of 75% of the administered dose in 24 h and 95% in 48 h.
  3-Methyl-Histidine was administered orally in 120 mg for one single dose, followed by a washout period of 1 week.
  Interventions: Dietary Supplement: 3-Methylhistidine
- Placebo (Placebo Comparator): Dextrose (glucose) was used in a dose of 20 g in this study.
  Interventions: Dietary Supplement: Amino Acid Supplement - One dose

INTERVENTIONS:
Dietary Supplement: Amino Acid Supplement - One dose — 20gr
  Arms: Arginine; Citrulline; Glutamine; Placebo
Dietary Supplement: 3-Methylhistidine — 120mgr
  Arms: 3-Methyl-Histidine

SUMMARY:
There are many forms of small bowel disease but their direct consequences on small bowel function are often very hard, if not impossible, to establish. It would be helpful if there was a reliable blood test to find out how well cells in the intestine are working. The amino acid citrulline is produced mainly by these cells, and therefore holds promise as a biological marker. Some previous studies have shown that fasting citrulline gave a good indication as to how many intestinal cells were present. However, other authors have not been able to confirm this.

Most of the citrulline in the blood is derived from another amino acid, glutamine, in a metabolic process that occurs in the intestinal cells, and most of the remainder comes from another amino acid, arginine. A further potential marker of intestinal cell function is the amino acid 3-methylhistidine. It is possible that a dynamic test, which incorporates time for conversion from one amino acid to another in the intestinal cells, might perform better.

The investigators therefore propose a study of oral glutamine, arginine, and 3-methylhistidine compared with citrulline itself or placebo (glucose) as it is hypothesized that these might increase the amount of citrulline more reproducibly. An initial study in healthy subjects is required to establish whether this is true, and if so to provide a normal range prior to investigation of patients who have or who might have the short bowel syndrome, and in whom the test would be clinically useful.

In this study, the subjects will take each of the amino acids and placebo in random order. Between each 6 hour-long visit the subjects will have at least one week where they are independent of the research team and during which they can behave normally. During each visit subjects will have a sequence of blood samples from an in-dwelling venous cannula, taken before and over 6 hours after a single small oral dose of that day's amino acid given as a small volume drink. Urine will also be collected for amino acid assay.

DETAILED DESCRIPTION:
Purpose and Design The purpose of the study is to determine the value of measuring citrulline after oral challenge, aiming to examine this as a function of enterocyte mass in patients with short bowel syndrome. The investigators hope to accumulate sufficient preliminary data in order to develop a new biochemical test for assessing absorption in future patient groups.

All subjects will provide written informed consent prior to their inclusion in the study. The study will be performed in accordance with International Conference on Harmonisation Guidelines for Good Clinical Practice (ICH GCP), the Helsinki Declaration and national regulations. Information about the study will be provided during one-on-one interviews with the help of a summary brochure which will be given to all potential subjects.

The study has been considered by the UK Medicines Agency, Medicines and Healthcare products Regulatory Agency (MHRA), and they agree that it is not a clinical trial of an investigational medicinal product.

Recruitment

1. Potential participants will be identified by the investigator's team. The sources will include hospital and investigator databases.
2. If permitted, advertisements will be posted for this study on University College London (UCL) electronic news sites, disseminated via UCL staff and student emails, with fliers to be posted on physical notice boards at UCL. Direct invitations from the researchers may also be attempted.
3. Healthy volunteers will be offered £7.85/hour for their participation in this study.

Consent Written informed consent will be obtained before any study-specific procedures are carried out.

All participants will be free to withdraw from the study at any time.

Risk, burdens and benefits Apart from the small risks associated with venous access the study is expected to be without important hazard. The agents to be administered are essentially constituents of the normal diet.

There is no expectation that participants will benefit from being in this study.

Confidentiality All data provided to the sponsor or designee will be identified only by subject number or initials, thereby ensuring that the subject's identity remains unknown.

What will happen at the end of the study? Participants will be given a summary of the key results and the opportunity for further discussion on request.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers fasted for at least 12 hours
2. Males and females aged at least 18

Exclusion Criteria:

1. Consumption of coffee or alcohol within 12 hours
2. Pregnancy
3. Use of any regular medication
4. Any significant past medical history

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-08; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve (AUC) for citrulline | predose, 15,30,45,60,90,120,180,360 minutes post-dose
  The primary end point for this study will be the Area Under the Curve (AUC) for citrulline after each oral load. This is the fraction of the administered dose that reaches the systemic circulation. Bioavailability is 100% for intravenous injection. It varies for other routes depending on incomplete absorption, first pass hepatic metabolism etc. Thus one plots plasma concentration against time, and the bioavailability is the AUC. The analysis of this continuous pharmacokinetic parameter will be performed on the plasma concentration-time data, using Statistical Package for the Social Sciences (SPSS) 17.0, Stata 10.0, Statistical Analysis System (SAS) and Sigma Plot.

CONTACTS AND LOCATIONS:
Overall Officials: Alastair Forbes, MD, FRCP, Principal Investigator — University College London, Centre for Gastroenterology
Locations (1):
- University College, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No